CLINICAL TRIAL: NCT00811200
Title: Treatment Of Radiation Retinopathy Trial Subtitle: Treatment of Radiation Retinopathy; Influence of Lucentis® and Kenalog® on Radiation Retinopathy After Irradiation of Choroidal Melanoma.
Brief Title: Treatment Of Radiation Retinopathy Trial
Acronym: TORR
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: M.J. Jager, MD, Phd, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P09.
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Uveal Melanoma
Keywords: radiation; retinopathy; maculopathy; choroidopathy; uveal; melanoma; lucentis; ranibizumab; kenalog; triamcinolone acetonide; radiation retinopathy after irradiation of uveal melanoma; radiation maculopathy after irradiation of uveal melanoma; radiation choroidopathy after irradiation of uveal melanoma
MeSH Terms: conditions — Uveal Melanoma; Retinal Diseases; Macular Degeneration; Choroid Diseases; Melanoma | interventions — Ranibizumab; Triamcinolone Acetonide; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1: Lucentis (Active Comparator)
  Interventions: Drug: ranibizumab
- 2: Kenalog (Active Comparator)
  Interventions: Drug: triamcinolone acetonide
- 3: No treatment (Sham Comparator)
  Interventions: Other: sham

INTERVENTIONS:
Drug: ranibizumab — three initial monthly intra vitreal injections with 0.5 mg ranibizumab
  Arms: 1: Lucentis
Drug: triamcinolone acetonide — at baseline one intra vitreal injection with 4.0 mg triamcinolone acetonide
  Arms: 2: Kenalog
Other: sham — at baseline one sham-injection
  Arms: 3: No treatment

SUMMARY:
The purpose of this study is to demonstrate a statistically significant improvement of visual acuity after treatment using either Lucentis® or Triamcinolone® compared to no treatment, in patients with radiation retinopathy.

DETAILED DESCRIPTION:
Approximately 30-40% of patients develop a deterioration of visual acuity within 5 years after treatment of uveal melanoma using radiation therapy and TTT due to radiation retinopathy (Shields 2002, Bartlema 2003). By administration of either Lucentis® or Triamcinolone® we hope to treat complications of radiation therapy, by demonstrating a statistically significant improvement in visual acuity and a reduced amount of macular edema and vascular leakage. Additionally, we hope to obtain a better understanding of the pathophysiologic processes involved, by demonstrating a possible relation between high levels of angiogenic factors (VEGF) in the anterior chamber fluid, and radiation retinopathy. In conclusion, we hope to provide evidence for a new therapy in patients with retinopathy, due to radiation in uveal melanoma. There is no scientifically proven treatment available at this time.

ELIGIBILITY:
Inclusion Criteria:

* The eye was previously irradiated for treatment of a uveal melanoma;
* Decrease of visual acuity after irradiation therapy by more than 10 letters (ETDRS) and is now 20/40 or less;
* Vision decrease is considered to be due to central radiation retinopathy with significant macular edema or optic disc edema;
* Age 18 years or older;
* The patient is fully competent;
* Written informed consent to participate in the trial is given.
* Patient is not pregnant (or not fertile) and is willing to use contraceptives for the duration of the trial (one year)
* Patient is willing and able to return for follow-up.

Exclusion Criteria:

* Vision decrease is considered to be due to ischemic radiation retinopathy without macular edema or optic disc edema;
* Other, approved therapy indicated for treatment of condition;
* Presence of metastasis;
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial;
* Pre-existing retinopathy due to other disorders;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
To demonstrate a statistically significant superiority of intravitreal ranibizumab (0.5mg) or triamcinolone acetonide (4.0mg) to no treatment, in the mean change from baseline in best corrected visual acuity (BCVA) | one year

SECONDARY OUTCOMES:
To evaluate the time course of BCVA changes on ranibizumab (0.5 mg) and triamcinolone acetonide (4.0mg) relative to no treatment. | one year
To evaluate the effects of ranibizumab (0.5 mg) and triamcinolone acetonide (4.0mg) on central retinal thickness, severity of retinopathy and other anatomical changes relative to no treatment | one year
To demonstrate a possible relation between decreasing levels of angiogenic factors (such as VEGF) in the anterior chamber fluid and a good response to treatment with ranibizumab or triamcinolone acetonide, and radiation retinopathy | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martine J Jager, MD, PhD, Principal Investigator — Leiden University Medical Center